CLINICAL TRIAL: NCT03753919
Title: A Phase II Study of Durvalumab (MEDI4736) Plus Tremelimumab for the Treatment of Patients with Progressive, Refractory Advanced Thyroid Carcinoma - the DUTHY Trial
Brief Title: Durvalumab Plus Tremelimumab for the Treatment of Patients with Progressive, Refractory Advanced Thyroid Carcinoma -The DUTHY Trial
Acronym: DUTHY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In compliance with current legislation applicable to Clinical Trials, following the instructions of the Spanish Agency for Medicines and Health Products.
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-T1812; 2018-001066-42 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Thyroid Papillary Carcinoma; Metastatic Thyroid Follicular Carcinoma; Metastatic Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: * Cohort 1: Advanced, radioiodine-refractory differentiated thyroid carcinoma, including papillary, follicular, Hürtle. Cell and poorly-differentiated thyroid carcinoma (DTC).
  * Cohort 2: Advanced medullary thyroid carcinoma (MTC).
  * Cohort 3: Advanced anaplastic thyroid cancer (ATC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab + Tremelimumab (Experimental): Durvalumab 1500 mg plus tremelimumab 75 mg every 4 weeks up to 4 cycles followed by durvalumab 1500 mg every 4 weeks until disease progression, unacceptable toxicity or patients' decision.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Subjects will be allocated in each primary tumor cohort to receive durvalumab 1500 mg every 4 weeks (Q4W) plus tremelimumab 75 mg Q4W for up to 4 doses during the first 4 cycles of combined therapy. After the first 4 cycles (or before is tremelimumab is stopped due to toxicity), patients will continue to receive durvalumab 1500 mg Q4W until disease progression or unacceptable toxicity. Cycles are defined by 4 weeks or 28 days.
  Other Names: MEDI4736
Drug: Tremelimumab — Subjects will be allocated in each primary tumor cohort to receive durvalumab 1500 mg every 4 weeks (Q4W) plus tremelimumab 75 mg Q4W for up to 4 doses during the first 4 cycles of combined therapy. After the first 4 cycles (or before is tremelimumab is stopped due to toxicity), patients will continue to receive durvalumab 1500 mg Q4W until disease progression or unacceptable toxicity. Cycles are defined by 4 weeks or 28 days.

SUMMARY:
This is a prospective, multi-centre, open label, stratified, exploratory phase II study evaluating the efficacy and safety of durvalumab plus tremelimumab in different cohorts of patients with thyroid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* Age ≥ 18 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Body weight >30kg.
* Confirmed differentiated thyroid cancer (papillary, follicular, poorly differentiated and Hürtle cell), medullary thyroid cancer and anaplastic thyroid cancer.
* Available tumor and blood samples for translational research
* Patients should meet one of the following criteria:

  1. Cohort 1: Patients with locally advanced or metastatic differentiated thyroid cancer (including the subtypes of papillary, follicular, poorly differentiated and Hürthle cell carcinoma) after disease progression on systemic therapy with MKIs. Patients could be recruited in the study after progression on Lenvatinib (regardless prior lines) or progression on at least two prior MKIs which may or not include Lenvatinib. No prior therapy with immune check point inhibitors is allowed. Patients with intolerable toxicity to MKIs that meet the prior inclusion criteria and experience disease progression by RECIST v1.1 after stopping therapy may be included.
  2. Cohort 2: Patients with locally advanced or metastatic medullary thyroid cancer after progression on systemic therapy with MKIs. Patients could be recruited in the study after progression to Vandetanib (regardless prior lines) or progression to at least two prior MKIs that may or not include Vandetanib. No prior therapy with immune check point inhibitors is allowed. Patients with intolerable toxicity to MKIs that meet the prior inclusion criteria and experience disease progression by RECIST v1.1 after stopping therapy may be included.
  3. Cohort 3: Patients with locally advanced or metastatic anaplastic thyroid cancer regardless of prior therapy. No prior therapy with immune check point inhibitors is allowed.
* No limitation of number of prior therapies.
* Life expectancy >3 months
* Adequate normal organ and marrow function as defined below: a) Haemoglobin ≥9.0 g/dL. b) Absolute neutrophil count (ANC) > 1500 per mm3. c) Platelet count ≥100,000 per mm3. d) Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician. e) AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal. f) Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre- menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: a) Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). b) Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 21 days.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Any previous treatment with a PD1, PD-L1 or CTLA-4 inhibitor, including durvalumab and tremelimumab.
* Any previous treatment with immunotherapy, including combinations of immunotherapy and other anticancer or targeted agents.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion: a) Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection). b) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent. c) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria: a) Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. b) Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: a) Patients with vitiligo or alopecia. b) Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement. c) Any chronic skin condition that does not require systemic therapy. d) Patients without active disease in the last 5 years may be included but only after consultation with the study physician. e) Patients with celiac disease controlled by diet alone.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of another primary malignancy except for: a) Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence. b) Adequately treated non-melanoma skin cancer or lentigomaligna without evidence of disease. c) Adequately treated carcinoma in situ without evidence of disease.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 90 days after the last dose of durvalumab monotherapy and 180 days for combined treatment with durvalumab and tremelimumab.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | 6 months
  Percentage of patients without progression of disease at month 6, according RECIST 1.1 criteria.
Overall survival rate at 6 months | 6 months
  Percentage of patients alive at month 6 from first dose of treatment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 42 months
  Response to treatment according to RECIST 1.1 criteria or iRECIST 1.1 criteria
Duration of response (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 42 months
  Length of time between start of treatment and date of evidenced response and progression of disease according irRECIST or RECIST 1.1 criteria, or death
Median progression-free survival | 42 months
  Length of time between date of evidenced response and progression of disease according irRECIST or RECIST 1.1 criteria, or death, or death
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 42 months
  Number and type of adverse events reported throughout the study period
Median Overall Survival | 42 months
  Length of time between start of treatment and death
Response status after start of study treatment | 6 and 12 months after start of the study treatment
  According irRECIST/RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, M.D., Ph.D., Study Chair — Hospital Universitari Vall d'Hebron, Barcelona
Locations (15):
- Spain (15):
  - Hospital Clínic Barcelona, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Instituto Catalán de Oncología de Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - MD Anderson Cancer Center, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Clínica Universidad de Navarra, Pamplona, Pamplona
  - Complejo Hospitalario Universitario de Vigo (CHUVI), Vigo, Spain
  - Hospital Provincial de Castellón, Castellon, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided